CLINICAL TRIAL: NCT07394595
Title: Upper Versus Lower Limb Cycling Exercise With Electrical Muscle Stimulation on Perceptual Responses, Energy Feelings in Young Adults
Brief Title: Upper Versus Lower Limb Cycling Exercise With Electrical Muscle Stimulation on Perceptual Responses, Energy Feelings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Assisstant professor, MTI University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB # 29/7/2024-2025
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Upper Limb Cycling with EMS (Experimental): Participants will perform cycling exercises using an arm ergometer combined with EMS applied to the upper limbs,Upper Limb Cycling with EMS: Participants will perform cycling exercises using an arm ergometer combined with EMS applied to the upper limbs. (Biceps, triceps, and deltoids) Jones et al., 2011
  Interventions: Other: Upper Limb Cycling with EMS
- Lower Limb Cycling with EMS (Experimental): Participants will engage in traditional cycling exercises using a stationary bike with EMS applied to the lower limbs,Lower Limb Cycling with EMS: Participants will engage in traditional cycling exercises using a stationary bike with EMS applied to the lower limbs. (Quadriceps, hamstrings, and calf muscles) Bax et al., 2005
  Interventions: Other: Lower Limb Cycling with EMS
- EMS upper and lower (Experimental): electrical stimulation upper and lower
  Interventions: Other: EMS upper and lower
- Control group (No Intervention): No exercises or intervention

INTERVENTIONS:
Other: Upper Limb Cycling with EMS — Upper Limb Cycling with EMS: Participants will perform cycling exercises using an arm ergometer combined with EMS applied to the upper limbs. (Biceps, triceps, and deltoids) Jones et al., 2011
  Arms: Upper Limb Cycling with EMS
Other: Lower Limb Cycling with EMS — Lower Limb Cycling with EMS: Participants will engage in traditional cycling exercises using a stationary bike with EMS applied to the lower limbs. (Quadriceps, hamstrings, and calf muscles)
  Arms: Lower Limb Cycling with EMS
Other: EMS upper and lower — EMS applied to the lower limbs. (Quadriceps, hamstrings, and calf muscles) and EMS applied to the upper limbs. (Biceps, triceps, and deltoids)
  Arms: EMS upper and lower

SUMMARY:
In comparing the two types of cycling exercises, the perceptual responses, such as perceived exertion and fatigue, as well as subjective feelings of energy, are crucial metrics. Lower limb cycling is traditionally associated with higher levels of exertion due to the larger muscle groups involved. However, when EMS is applied, both upper and lower limb cycling might exhibit altered perceptions of effort and energy levels, with EMS potentially equalizing the exertional differences. This research is significant for designing exercise programs that optimize energy expenditure and enhance performance, particularly in rehabilitative settings or for individuals looking to diversify their physical training regimens.

DETAILED DESCRIPTION:
Perceptual responses, such as perceived exertion and enjoyment, play a critical role in exercise adherence and overall experience. By examining the differences in these responses between upper and lower limb cycling combined with EMS, we can identify which modality might be more favorable for maintaining motivation and engagement in young adults. This demographic is particularly crucial as they transition into lifelong fitness habits. Exploring how EMS impacts these perceptual responses can provide insights into optimizing exercise regimens for enhanced user experiences, potentially leading to better adherence and improved fitness outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-45 years
* No history of cardiovascular or musculoskeletal disorders
* Physically active individuals with a minimum of 150 minutes of moderate exercise per week

Exclusion Criteria:

* Current use of medications affecting muscle function
* Pregnant or lactating individuals
* Involvement in other structured exercise programs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Perceptual Responses | at baseline and at 8 weeks
  Assessed using the Rate of Perceived Exertion (RPE) scale.
Self-Perceived Energy Feeling | at baseline and at 8 weeks
  (All participants will fill a short questionnaire (from 1 to 5 points) about their perception of energy before every training. Energy Feeling will be assessed (Evergy level, Fatigue Level, Feeling of Alertness, and Feeling of Focus for the task, valued from 1 = low energy to 5 = high energy).

SECONDARY OUTCOMES:
Perception of Effort during Endurance Training | at baseline and at 8 weeks
  (Borg Scale (6-20) will be used to collect the perception of effort during endurance training (every 5 minutes) and 15-20 minutes after each session).
Blood lactate concentration | at baseline and at 8 weeks
  measured using capillary puncture during submaximal and maximal incremental exercise

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy ,Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No